CLINICAL TRIAL: NCT05697341
Title: A Comparative Study Between Ultra Mini Percutaneous Nephrolithotomy Versus Stented Extracorporeal Shock Wave Lithotripsy for Treatment of Renal Stones in Egypt
Brief Title: Ultra Mini Percutaneous Nephrolithotomy VS Stented Extracorporeal Shock Wave Lithotripsy for Stone Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Younan Ramsis Samir, Lecturer of Urology, Faculty of medicine, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YRS0001
Record Dates: First submitted 2023-01-13; First posted 2023-01-25 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Renal Stone
Keywords: Nephrolithiasis; Ultra-Mini-PCNL; Stented SWL
MeSH Terms: conditions — Nephrolithiasis

STUDY DESIGN:
Intervention Model Description: 90 Patients were enrolled from the outpatient urology clinic of Ain Shams University hospital (Demredash Hospital) randomized to either Group A Ultra-Mini-Percutaneous nephrolithotomy group or Group B stented SWL group via the closed envelope method.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultra-Mini-PCNL Group (A) (Active Comparator): In The Ultra-Mini-percutaneous nephrolithotomy group, a 5 Fr open-ended ureteral catheter was introduced and a retrograde pyelogram was performed in the Lithotomy position after the induction of general anesthesia. Patients were then repositioned to the prone position. Ultra-mini-PCNLs were done in a prone position by a single consultant. The desired calyx was punctured with a Cook diamond tip 18G puncture needle under fluoroscopy guidance using standard bull's eye technique. Single tract dilatation with One Step Dilator (11Fr), with central channel for guide wires with its Operating Sheath (Storzz Dilator and Operating Sheaths for MIP XS) under fluoroscopy guidance. Storzz Nephroscope for MIP XS / S along with Swiss Lithoclast master pneumatic lithotripter with 1/0.8 mm probe was used for stone fragmentation. Stone fragments are flushed out on rapid removal of the endoscope, due to a 'vortex' effect and with wash through the operating sheath using a 6 Fr. nelaton catheter.
  Interventions: Procedure: Ultra-Mini-PCNL
- Stented SWL Group (B) (Active Comparator): In the stented ESWL group, a 5 Fr open-ended ureteral catheter was introduced in the renal pelvis, and a retrograde pyelogram was performed in the Lithotomy position after the induction of general anathesia. JJ is applied either 5-26 or 5-28 accorging to the patient. Extracorporeal shock wave lithotripsy ESWL was administered with an electromagnetic shockwave lithotripter (Siemens electromagnetic lithotripters devices). Patients were positioned supine with the shock head from the back. Fluoroscopy was used for the localization and monitoring of stone fragmentation. All patients received shocks at a frequency of 60/min. An average of approximately 2500-3000 shocks was targeted in all patients.
  Interventions: Procedure: Stented SWL

INTERVENTIONS:
Procedure: Ultra-Mini-PCNL — treatment to extract or disintegrate renal stones
  Arms: Ultra-Mini-PCNL Group (A)
Procedure: Stented SWL — treatment to disintegrate renal stones in the presence of a JJ
  Arms: Stented SWL Group (B)

SUMMARY:
Nephrolithiasis is the third most common disease of the urinary tract. As minimally invasive technologies develop, shock wave lithotripsy (SWL), retrograde intrarenal surgery (RIRS), and percutaneous nephrolithotomy (PCNL) are different surgeries to treat renal stones.

Aim of the Study is to compare results, safety and outcome of Ultra mini PCNL versus stented extracorporeal shock wave lithotripsy (SWL) for the management of renal calculi from 10 - 20 mm. Patients were randomized to either Ultra-Mini-Percutaneous nephrolithotomy group or stented SWL group via the closed envelope method. Patient data was collected preoperatively, immediately postoperatively and 2 and 4 weeks postoperatively to assess operative time, hospital stay, complications regarding fever, hematuria and need for blood transfusion, residual stones and need for retreatment.

DETAILED DESCRIPTION:
Nephrolithiasis is the third most common disease of the urinary tract, following urinary tract infections and Prostatic diseases. It also has a 1-year recurrence rate of 7% and 10-year recurrence rate of 50%.

Management of renal stones had seen a great shift over the last ten years. The need to find a balance between morbidity and stone clearance is always the milestone of treatment choice. Low risk procedure with high retreatment percentage vs another relatively higher risk procedure with lower retreatment chances.

As minimally invasive technologies develop, shock wave lithotripsy (SWL), retrograde intrarenal surgery (RIRS), and percutaneous nephrolithotomy (PCNL) are different surgeries to treat renal stones. Open, laparoscopic, and robotic surgeries have their place only in highly selected patients.

In the European Association of Urology (EAU) Guidelines on Urolithiasis, PCNL is a treatment of choice (TOC) for renal stones > 20 mm, SWL or RIRS is the first-line therapy for renal stones < 10 mm, and SWL or endourologic treatment (all PCNL and ureteroscopic interventions) can be performed for stones 10-20 mm.

SWL is a minimally invasive intervention with good patient tolerance; it is regarded as the first line treatment for nephrolithiasis < 20 mm in size. Poor clearance of lower calyceal stone fragments due to gravity or unfavorable infundibulopelvic angle limits the efficacy of SWL for treating lower calyceal stones.

flexible ureteroscopy increased quality and performance of upper urinary tract exploration, allowing the treatment the majority of stones at all sites. Experiences with RIRS have revealed higher stone-free rate (SFR) with less risk of renal damage and bleeding. Nevertheless, RIRS is also associated with some disadvantages as the possible need for staged procedures, risk of ureteral injuries and the costs of acquisition and maintenance of the complex endourological instruments and those issues can be possible factors that might have limited the capillary diffusion of this endoscopic procedure.

Percutaneous nephrolithotripsy (24-30F) remains the standard procedure for treating large renal calculi. While achieving high SFR, it also has many drawbacks such as bleeding, postoperative pain, and a long recovery period due to its large access tract, so the mini percutaneous nephrolithotripsy (14-22F) with a smaller tract size came into existence. To reduce renal parenchymal injury associated with standard PCNL, minimally invasive PCNL with a smaller tract size has been developed. Depending on the size of the access tract, minimally invasive PCNL can be classified into Mini-PCNL (14- 22Fr), Ultra-mini-PCNL (11-13Fr).

PCNL carried a significantly higher stone free rate than RIRS, especially for lower calyceal stones (OR=2.65, P=.003), however Mini-PCNL was at the expense of a longer hospital stay and an increased hemoglobin drop.

Although PCNL could exhibit a stone free rate of 93.8%, a global survey revealed that it carried a complication rate of up to 14.5%.

Ulra-mini-PCNL offer a particular advantage for difficult to access calculi, impacted lower pole calculi with an acute infundibular angle or stones in a calyceal diverticulum, with the greater advantage of reduced bleeding.

This study was conducted at Urology department, Faculty of Medicine, Ain Shams University. Inclusion criteria included patients between 18 and 60 years, complaining of radioopaque renal stones ranging from 10-20 mm with BMI not exceeding 40 Exclusion criteria were patients who had radiolucent stones, smaller than 10 mm or larger than 20 mm, with congenital renal anomalies or spinal deformity or BMI exceeding 40. Patients with uncorrected bleeding diathesis or pregnant females or untreated urinary tract infection were also excluded.

In this study patients were recruited from the outpatient urology clinic between March 2021 till March 2022.

Using Power Analysis and Sample Size Software version 15 program for sample size calculation after reviewing results from a previous study (Zhang et al, 2019) we assume a medium effect size difference between the two groups regarding the stone-free rate ( d=0.6), based on these findings sample size of 90 patients (45 per group) achieve 80% power to reject the null hypothesis of zero effect size when the population effect size is 0.60 and the significance level (alpha) is 0.050 using a two-sided z test.

Patients were randomized to either Group A Ultra-Mini-Percutaneous nephrolithotomy group or Group B stented SWL group via the closed envelope method.

Preoperative evaluation including careful history taking, general and local examination, urine analysis, perioperative labs (CBC, bleeding profile, liver and renal functions), Computerized tomography Urinary Tract (CTUT) with Hounsfield unit estimation and Plain X-ray of the urinary tract (KUB).

All patients were given perioperative antibiotic prophylaxis. In The Ultra-Mini-percutaneous nephrolithotomy group, a 5 Fr open-ended ureteral catheter was introduced in the renal pelvis, and a retrograde pyelogram was performed in the Lithotomy position after the induction of general anesthesia. Patients were then repositioned to the prone position. Ultra-mini-PCNLs were done in a prone position by a single consultant. The desired calyx was punctured with a Cook diamond tip puncture needle under fluoroscopy guidance using standard bull's eye technique. Single tract dilatation with One Step Dilator (11Fr), with central channel for guide wires with its Operating Sheath (Storz Dilator and Operating Sheaths for Minimal Invasive PCNL (MIP) XS) under fluoroscopy guidance. Storz Nephroscope for MIP XS / S along with Swiss Lithoclast master pneumatic lithotripter with 1/0.8 mm probe was used for stone fragmentation. Stone fragments are flushed out on rapid removal of the endoscope, due to a 'vortex' effect and with wash through the operating sheath using a 6 Fr. nelaton catheter.

In the stented Extracorporeal ShockWave Lithotripsy (ESWL) group, a 5 Fr open-ended ureteral catheter was introduced in the renal pelvis, and a retrograde pyelogram was performed in the Lithotomy position after the induction of general anaesthesia JJ is applied either 5-26 or 5-28 according to the patient. ESWL was administered with an electromagnetic shockwave lithotripter (Siemens electromagnetic lithotripters devices). Patients were positioned supine with the shock head from the back. Fluoroscopy was used for the localization and monitoring of stone fragmentation. All patients received shocks at a frequency of 60/min. An average of approximately 2500-3000 shocks was targeted in all patients.

Follow up of patients was done postoperative immediately including careful and detailed history taking and examination including pain, fever, sepsis, and hematuria. Serum Hb level, S.creatinine, BUN, Na+, K+

ELIGIBILITY:
Inclusion Criteria:

* patients between 18 and 60 years
* complaining of radioopaque renal stones ranging from 10-20 mm.
* BMI not exceeding 40

Exclusion Criteria:

* radiolucent stones,
* smaller than 10 mm or larger than 20 mm stones
* congenital renal anomalies or spinal deformity
* BMI exceeding 40.
* Patients with uncorrected bleeding diathesis
* pregnant females
* untreated UTI.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Stone-free status | at 2 or 4 weeks after ultra-mini-PCNL or stented SWL
  The complete stone clearance or presence of clinically insignificant residual fragments (<4 mm) 2 or 4 weeks after the final procedure was regarded as stone-free

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Radwan, MD, Study Chair — Assisstant Professof of Urology, Faculty of medicine, Ain Shams University
Locations (1):
- Ain Shams University, Faculty of medicine, Cairo, Abbassia, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Skolarikos A, Straub M, Knoll T, Sarica K, Seitz C, Petrik A, Turk C. Metabolic evaluation and recurrence prevention for urinary stone patients: EAU guidelines. Eur Urol. 2015 Apr;67(4):750-63. doi: 10.1016/j.eururo.2014.10.029. Epub 2014 Nov 20. PMID 25454613
- [Background] Kim CH, Chung DY, Rha KH, Lee JY, Lee SH. Effectiveness of Percutaneous Nephrolithotomy, Retrograde Intrarenal Surgery, and Extracorporeal Shock Wave Lithotripsy for Treatment of Renal Stones: A Systematic Review and Meta-Analysis. Medicina (Kaunas). 2020 Dec 30;57(1):26. doi: 10.3390/medicina57010026. PMID 33396839
- [Background] Gao XS, Liao BH, Chen YT, Feng SJ, Gao R, Luo DY, Liu JM, Wang KJ. Different Tract Sizes of Miniaturized Percutaneous Nephrolithotomy Versus Retrograde Intrarenal Surgery: A Systematic Review and Meta-Analysis. J Endourol. 2017 Nov;31(11):1101-1110. doi: 10.1089/end.2017.0547. Epub 2017 Oct 30. PMID 28950716
- [Background] Bozzini G, Verze P, Arcaniolo D, Dal Piaz O, Buffi NM, Guazzoni G, Provenzano M, Osmolorskij B, Sanguedolce F, Montanari E, Macchione N, Pummer K, Mirone V, De Sio M, Taverna G. A prospective randomized comparison among SWL, PCNL and RIRS for lower calyceal stones less than 2 cm: a multicenter experience : A better understanding on the treatment options for lower pole stones. World J Urol. 2017 Dec;35(12):1967-1975. doi: 10.1007/s00345-017-2084-7. Epub 2017 Sep 5. PMID 28875295